CLINICAL TRIAL: NCT00410059
Title: A Phase II, Open Label Study of Erlotinib (Tarceva) in Previously Treated Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: BATTLE Program: Erlotinib in Previously Treated Subjects With Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0824; NCI-2012-02083 (Registry Identifier: NCI CTRP); W81XWH-06-1-0303 (Other: DOD)
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; NSCLC; Erlotinib; Tarceva; OSI-774; Battle Program
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental): Erlotinib 150 mg by mouth daily x 28 days.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — 150 mg by mouth daily x 28 days
  Other Names: Tarceva; OSI-774; Erlotinib Hydrochloride

SUMMARY:
The goal of this clinical research study is to learn if erlotinib hydrochloride (OSI-774, Tarceva®) can help to control NSCLC. The safety of this drug will also be studied, as well as the drug's effect on different cells in the body and the participants' overall response.

DETAILED DESCRIPTION:
Erlotinib hydrochloride is designed to block the activity of an enzyme found on the surface of many tumor cells that may slow tumor growth.

In order to enroll in this study, you must also be enrolled in Protocol 2005-0823: A Biomarker-integrated study in Chemorefractory Patients with Advanced Non-Small Cell Lung Cancer. Protocol 2005-0823 is the screening study in a group of studies called the BATTLE program. Participants in Protocol 2005-0823 are assigned to one of the research studies. The results of your tumor analysis helped the study doctor determine to assign you to this particular research study.

While on study, you will take erlotinib hydrochloride by mouth once a day. Tablets should be taken preferably in the morning 1 hour before or 2 hours after a meal with no more than 7 ounces of water. If you are unable to swallow tablets, you may dissolve the tablets in distilled water. If you forget to take a dose, the last missed dose should be taken as soon as you remember, as long as it is at least 12 hours before the next dose is due to be taken. The next day, you should take the scheduled dose at the usual time. Every attempt should be made to keep from vomiting the medication for at least 30 minutes after taking it. For example, if you feel nauseated before or after taking the erlotinib, anti-nausea medications should be used. The dose of erlotinib hydrochloride may be repeated if vomiting occurs within 30 minutes of taking the tablet. Four (4) weeks is considered 1 treatment cycle.

Every 4 weeks, your complete medical history will be recorded and you will have a physical exam, including measurement of vital signs (blood pressure, pulse, temperature, breathing rate) and weight. You will have blood drawn (about 2 teaspoons) for routine tests. You will have a performance status evaluation (questions about your ability to perform everyday activities). Your study doctor will ask you about any medications you are taking and your smoking history. Every 2 cycles, the tumor will be evaluated by chest x-ray and computed tomography (CT) or magnetic resonance imaging (MRI) scans to evaluate the status of the disease. If you are taking warfarin, you will have blood drawn (about 1-2 teaspoons) to check your blood clotting function weekly for the first 5 weeks of treatment and then every cycle after that.

You may continue receiving erlotinib hydrochloride for as long as the cancer responds to study treatment. Your doctor may decide to take you off this study if you experience intolerable side effects, your medical condition gets worse, or you are unable to comply with study requirements. If you stop study treatment, you may be able to enroll in 1 of the remaining 3 protocols of the BATTLE program. You should discuss this with your doctor.

After you have stopped taking the study treatment, you will have a physical exam, including measurement of vital signs. Blood (about 2 teaspoons) and urine will be collected for routine tests. You will also have blood drawn (about 1-2 teaspoons) to check your blood clotting function. You will have a performance status evaluation, a chest x-ray, and a CT or MRI scan. Following this evaluation, you will be contacted by telephone every 3 months for up to 3 years, to see how you are doing.

You have the right to leave the study at any time. If you choose to stop participating in this study, you should contact the study chair and/or research nurse. Your doctor may decide to take you off this study if your medical condition gets worse and/or you are unable to comply with study requirements.

This is an investigational study. Erlotinib hydrochloride is approved by the FDA for treatment of NSCLC in patients who have relapsed. Up to 72 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration.
2. The patient has a diagnosis of either stage IIIB, stage IV, or advanced, incurable NSCLC, and failed at least one front-line metastatic NSCLC chemotherapy regimen. (Patients who have failed adjuvant or locally advanced therapy within 6 months are also eligible to participate in study).
3. The patient has uni-dimensionally measurable NSCLC.
4. Karnofsky performance status >/= 60 or ECOG performance status 0-2
5. The patient has biopsy accessible tumor.
6. The patient has adequate hematologic function as defined by an absolute neutrophil count (ANC) >/= 1,500/mm^3, platelet count >/= 100,000/mm^3, WBC >/= 3,000/ mm^3, and hemoglobin >/= 9 g/dL.
7. The patient has adequate hepatic function as defined by a total bilirubin level </= 1.5 X the upper limit of normal, and alkaline phosphatase, AST or ALT </= 2.5 X the upper limit of normal.
8. The patient has adequate renal function as defined by a serum creatinine level </= 1.5 mg/dL or a calculated creatinine clearance of >/= 60cc/minute.
9. The patient has PT < 1.5 x upper limit of normal
10. If patient has brain metastasis, they must have been stable (treated or asymptomatic) for at least 4 weeks after radiation, if treated with radiation, and not have used steroids for at least 1 week. Re-imaging performed after 2 weeks, upon completion of radiation therapy.
11. The patient is >/= 18 years of age.
12. The patient has signed informed consent.
13. The patient is eligible if disease free from a previously treated malignancy, other than a previous NSCLC, for greater than two years. Patients with a history of prior basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix are exempt from exclusion.
14. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of tudy participation. Childbearing potential will be defined as women who have had menses within the past 12 months,who have not had tubal ligation or bilateral oophorectomy.Should a woman become pregnant or suspect that she is pregnant while participating in this study,she should inform her treating physician immediately.The patient,if a man,agrees to use effective contraception or abstinence.
15. Subject must be considered legally capable of providing his or her own consent for participation in this study.

Exclusion Criteria:

1. The patient has received prior investigational therapy, chemotherapy, surgery, or radiotherapy within 4 weeks of initiating study drug
2. The patient has undergone prior thoracic or abdominal surgery within 28 days of study entry, excluding prior diagnostic biopsy.
3. The patient has received radiation therapy to the measurable tumor within 6 months. Patients are allowed to have local irradiation for the management of tumor-related symptoms (bones, brain). However, if a patient has active new disease growing in the previously irradiated site, the patient will be eligible to participate in the study.
4. The patient has a significant medical history or unstable medical condition (unstable systemic disease: congestive heart failure (New York Heart Association Functional Classification class II or worse), recent myocardial infarction within 3 months, unstable angina, active infection (i.e. currently treated with antibiotics, uncontrolled hypertension). Patients with controlled diabetes will be allowed. Patient must be able to undergo procedure for tissue acquisition.
5. The patient has uncontrolled seizure disorder, active neurologic disease, or neuropathy >/= grade 2. Patients with meningeal or CNS involvement by tumor are eligible for the study if the above exclusion criteria are not met.
6. The patient is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding.
7. Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment.
8. The patient is actively taking herbal remedies or over-the-counter biologics (e.g., shark cartilage, high dose antioxidants).
9. Patients will be allowed to have prior biologic (i.e. VEGF, EGFR, etc.) therapy. However, the patient will be excluded from a given study if he/she has received the same therapy as the clinical trial (i.e. If a patient has been previously treated with bevacizumab, they are allowed to enroll in any of the 4 studies. If a patient has been previously treated with erlotinib, they are excluded from the clinical trials with erlotinib). In addition, if a patient has been previously treated with gefitinib (Iressa), they are excluded from the clinical trials with erlotinib.
10. The patient has dysphagia. A patient who is unable to swallow intact capsules must be able to swallow capsules dissolved in water.
11. The patient has active gastrointestinal disease or a disorder that alters gastrointestinal motility or absorption (i.e., lack of integrity of the gastrointestinal tract such as a significant surgical resection of the stomach or small bowel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erminia Massarelli, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gong K, Guo G, Beckley N, Zhang Y, Yang X, Sharma M, Habib AA. Tumor necrosis factor in lung cancer: Complex roles in biology and resistance to treatment. Neoplasia. 2021 Feb;23(2):189-196. doi: 10.1016/j.neo.2020.12.006. Epub 2020 Dec 26. PMID 33373873
- [Derived] Tam AL, Kim ES, Lee JJ, Ensor JE, Hicks ME, Tang X, Blumenschein GR, Alden CM, Erasmus JJ, Tsao A, Lippman SM, Hong WK, Wistuba II, Gupta S. Feasibility of image-guided transthoracic core-needle biopsy in the BATTLE lung trial. J Thorac Oncol. 2013 Apr;8(4):436-42. doi: 10.1097/JTO.0b013e318287c91e. PMID 23442309
- [Derived] Kim ES, Herbst RS, Wistuba II, Lee JJ, Blumenschein GR Jr, Tsao A, Stewart DJ, Hicks ME, Erasmus J Jr, Gupta S, Alden CM, Liu S, Tang X, Khuri FR, Tran HT, Johnson BE, Heymach JV, Mao L, Fossella F, Kies MS, Papadimitrakopoulou V, Davis SE, Lippman SM, Hong WK. The BATTLE trial: personalizing therapy for lung cancer. Cancer Discov. 2011 Jun;1(1):44-53. doi: 10.1158/2159-8274.CD-10-0010. Epub 2011 Jun 1. PMID 22586319
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 29, 2006 to February 4, 2010. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Erlotinib: 150 mg orally day for 28 days.
Period: Overall Study
Arm/Group | Erlotinib
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: 8 Week Progression-Free Survival Rate (i.e. Disease Control Rate)
Description: Progression-free survival (i.e. disease control rate) defined as percentage of participants without progression at 8 weeks, evaluation after the second cycle of therapy (i.e., 8 weeks), with confirmation of efficacy 2 cycles after its initial assessment. A "success" or "disease control" to treatment is defined as a participant being progression free at 8 weeks after randomization.
Time Frame: Radiographic evaluation after cycle 2 (8 weeks of therapy)
Population: One participant was not evaluable for outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 58
Participants | 20

ADVERSE EVENTS:
Time Frame: Adverse event data collected over two cycles (28-day cycle) up to 60 days.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 1/59
Other Adverse Events (participants affected / at risk) | 57/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=59)
Melena (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=59)
Acne (Skin and subcutaneous tissue disorders) | 17 (18)
Diarrhea (Gastrointestinal disorders) | 16 (21)
Fatigue (Gastrointestinal disorders) | 9 (13)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 15 (16)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Bilirubin Increase (Investigations) | 3 (3)
Dry Eyes (Eye disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nail Changes (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7)
Pain (other) (General disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 16 (16)
Weight Loss (Investigations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes